CLINICAL TRIAL: NCT05737186
Title: The Efficacy and Safety of SGLT2 Inhibitors in Improving Heart Failure in Patients With Chronic Heart Failure With Reduced Ejection Fraction (HFrEF) and Severe Renal Insufficiency
Brief Title: SGLT2 Inhibitors and Treatment of Heart Failure in Severe Renal Insufficiency
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Double blind packaged drug is up to expiration date
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Ren qian, Associate Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAPA-FF
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Drug: SGLT-2 inhibitor
- Control group (No Intervention)

INTERVENTIONS:
Drug: SGLT-2 inhibitor — dapagliflozin
  Arms: Intervention group

SUMMARY:
In the treatment of heart failure (HF), SGLT-2 inhibitor (SGLT-2i) can significantly improve the clinical outcome and quality of life related to HF. The current data show that SGLT-2i is effective and safe in improving HF outcomes in patients with chronic kidney disease (CKD) stage 4, but there is little clinical evidence in patients with eGFR<20 ml/min/1.73 m2. Therefore, our research is designed to confirm that SGLT-2i can improve the outcome of HF in patients with chronic heart failure with reduced ejection fraction (HFrEF) and severe chronic renal insufficiency (eGFR<20ml/min/1.73m2).

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years
* Patients with clinically confirmed chronic heart failure who have received treatment for heart failure according to the guidelines in the past two months, New York Heart Association (NYHA) grade II-IV
* Left ventricular ejection fraction (LVEF) ≤ 40% in the past 1 year
* Clinically confirmed chronic renal insufficiency, eGFR<20ml/min/1.73m2 or maintenance hemodialysis

Exclusion Criteria:

* Allergy to SGLT-2i
* ALT or AST >3 times the upper limit of normal value; Or total bilirubin>2 times the upper limit of normal value
* Urinary or reproductive system infection in the last month
* Blood potassium is greater than or equal to the upper limit of normal value
* Patients with acute heart failure
* Patients who need intravenous diuretics before randomization, and the dose is greater than 40mg furosemide, or other equivalent intravenous loop diuretics
* Patients who need intravenous vasodilators, including nitrates, before randomization
* Systolic blood pressure<100mmHg measured during screening or at randomization
* Hemoglobin<90g/L
* Uncontrolled serious arrhythmia
* Myocardial infarction, unstable angina pectoris, hemorrhagic stroke or ischemic stroke in 90 days before randomization
* Proliferative retinopathy or macular disease, painful diabetes neuropathy, diabetes foot, diabetes ketoacidosis, hyperglycemic hyperosmolality that needed treatment in 90 days before randomization
* Patients with malignant tumors
* Drug or alcohol addicts
* Patients who have donated or transfused blood within 90 days before randomization, or are expected to donate or transfuse blood during the study period
* Pregnant or lactating women, or patients who cannot take reliable contraceptive measures during the study period
* Patients with uncontrolled abnormal thyroid function
* Type 1 diabetes
* Not suitable evaluated by the investigator

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
The quality of Life | 12 weeks
  The change of Quality of Life in patients by using the The Kansas City Cardiomyopathy Questionnaire(KCCQ)

SECONDARY OUTCOMES:
The quality of Life | 2 weeks, 4weeks and 8weeks
  The change of Quality of Life in patients by using the KCCQ
Dose changes of diuretics | 12 weeks
  Dose changes of diuretics in subgroups of patients without dialysis
Changes of eGFR | 2 and 12 weeks
  Changes of eGFR in the subgroup of non-dialysis patients at 2 and 12 weeks
Changes of brain natriuretic peptide (BNP) | 12 weeks
  Changes of BNP
Changes of body weight | 12 weeks
  Changes of Body weight and BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Please Select, China